CLINICAL TRIAL: NCT00637559
Title: A Multicenter, Double-blind, Three-way Crossover Intraesophageal and Intragastric pH Study of Three Esomeprazole Treatment Regimens in Documented Barrett's Esophagus Patients
Brief Title: Barrett's Esophagus - 315 - 3 Way Cross-Over
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, Astra Zeneca
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 315; D9612L00056
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Barrett's Esophagus
Keywords: Nexium; Barrett's esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Esomeprazole

ARMS (3):
- 1 (Experimental): 40mg twice daily
  Interventions: Drug: Esomeprazole Magnesium
- 2 (Experimental): 40mg three times daily
  Interventions: Drug: Esomeprazole Magnesium
- 3 (Experimental): 20mg three times daily
  Interventions: Drug: Esomeprazole Magnesium

INTERVENTIONS:
Drug: Esomeprazole Magnesium
  Other Names: Nexium

SUMMARY:
This study looks the intragastric and intraesophageal pH in patients with documented Barrett's esophagus whilst taking esomeprazole 40mg twice daily, esomeprazole 40mg three times daily, esomeprazole 20 mg three times daily.

ELIGIBILITY:
Inclusion Criteria:

* Must have a previously established, biopsy-proven diagnosis of Barrett's esophagus with segment length greater than 3cm, with no dysplasia or adenocarcinoma within the previous 12 months

Exclusion Criteria:

* A history of esophageal, gastric, or duodenal surgery, including anti-reflux surgery or endoscopic anti-reflux procedures, except for simple closure of a gastric or duodenal ulcer.
* History of various gastrointestinal diseases - please see investigator for full list.
* Evidence of any malignant disease in the last 5 years, except minor superficial skin disease.
* Unstable diabetes mellitus. Stable on a controlled diet, oral agents or insulin are acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2002-03; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
To compare the total percent time during the 24-hour monitoring period that gastric pH is above 4.0 at steady state in patients when taking: esomeprazole 40mg twice daily, esomeprazole 40mg three times daily, esomeprazole 20 mg three times daily. | pH measured on Day 5

SECONDARY OUTCOMES:
Compare total percent time distal esophageal pH is above 4.0 at steady state for each treatment period. | pH measured

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca